CLINICAL TRIAL: NCT01502137
Title: An Open, Non-randomized, Single-centre, Parallel Group Trial Investigating the Steady-state Blood Concentration Profile and Effects of Once Daily Subcutaneously Injected Recombinant Human Growth Hormone (Norditropin® SimpleXx®) in Patients With End Stage Renal Disease Receiving Chronic Haemodialysis and in Matched Healthy Subjects
Brief Title: Pharmacokinetics of Somatropin in Patients With End Stage Renal Disease Receiving Chronic Haemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1630-1559; 2005-000765-19 (EudraCT Number)
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Kidney Disease; End-Stage Renal Disease; Healthy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESRD patients (Experimental)
  Interventions: Drug: somatropin
- Healthy subjects (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Injected subcutaneously, 50 mcg/kg/day (up to a maximum of 4 mg/day) once daily. Additional dose administered during dialysis. In total, patients will receive 8 doses.
  Arms: ESRD patients
Drug: somatropin — Injected subcutaneously, 50 mcg/kg/day (up to a maximum of 4 mg/day) once daily. Additional dose administered during dialysis. In total, subjects will receive 7 doses.
  Arms: Healthy subjects

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to to compare steady-state total growth hormone (GH) exposure in haemodialysis (HD) patients with that of matched healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS:
* Male or female, age equal to or above 18 years undergoing chronic haemodialysis
* Stable and adequate haemodialysis treatment three months prior to enrolment
* HEALTHY SUBJECTS:
* Matching an individual of the patient group by: Gender and age (± 5 years)
* Matching an individual of the patient group by weight (after dialysis, ±10%)
* Creatinine clearance above 80 ml/min
* Subjects must be in good health in accordance with their age as determined by a medical
* history, physical examination, vital signs, ECG (electrocardiogram), routine haematology and clinical chemistry

Exclusion Criteria:

* Use of cuprophane membranes
* Active malignant disease
* Diabetes
* Critical illness as defined by the need of respiratory or circulatory support
* Known or suspected allergy to the trial product
* Pregnancy, breast feeding, the intention of becoming pregnant or fertile women judged to be
* using inadequate contraceptive measures
* Blood Pressure (pre-dialysis) above 180/110
* Chronic treatment with steroids in doses above 10 mg/day prednisolone (or equivalent)
* Treated with immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-06; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Growth hormone exposure at steady state

SECONDARY OUTCOMES:
Area under the Curve (AUC)
t½ (terminal half-life)
Cmax (maximum plasma concentration)
tmax (time to reach maximum)
IGF-I (Insulin-Like Growth Factor I)
Adverse events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, München, Germany

REFERENCES:
- [Result] Langbakke IH, Nielsen JN, Skettrup MP, Harper A, Klitgaard T, Weil A, Engelhardt E, Lange M. Pharmacokinetics and pharmacodynamics of growth hormone in patients on chronic haemodialysis compared with matched healthy subjects: an open, nonrandomized, parallel-group trial. Clin Endocrinol (Oxf). 2007 Nov;67(5):776-83. doi: 10.1111/j.1365-2265.2007.02962.x. Epub 2007 Jul 18. PMID 17634080
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com